CLINICAL TRIAL: NCT01447992
Title: Pilot Study 1 of Outpatient Control-to-Range - System and Monitoring Testing
Brief Title: Feasibility Study of a Portable Artificial Pancreas System in Type 1 Diabetes Mellitus (T1DM) - Padova
Acronym: HomeCTR1_2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Padova (Other); University Hospital, Montpellier (Other); University of California, Santa Barbara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2433P; JDRF 22-2011-649 (Other Grant/Funding Number: Juvenile Diabetes Research Foundation)
Record Dates: First submitted 2011-09-29; First posted 2011-10-06 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas; Insulin Pump; Continuous Glucose Monitor; Closed Loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Portable artificial pancreas system with Control-To-Range (Experimental)
  Interventions: Device: Portable artificial pancreas system with Control-To-Range

INTERVENTIONS:
Device: Portable artificial pancreas system with Control-To-Range — We will test the new portable Control-To-Range system in clinical research center conditions for 10 hours followed by 18 hours of Control-To-Range in a hotel.

SUMMARY:
A single arm, single treatment study is proposed to assess the feasibility of a portable artificial pancreas system outside of a hospital based clinical research center.

Adult T1DM patients will use a newly developed platform in conjunction with a subcutaneous insulin infusion pump and a continuous glucose monitor for 18 hours is quasi free conditions (hotel).

DETAILED DESCRIPTION:
Automated closed-loop control (CLC), known as "artificial pancreas" (AP) can have tremendous impact on the health and lives of people with type 1 diabetes (T1D). Our inter-institutional and international research team has been on the forefront of CLC developments since the beginning of the Juvenile Diabetes Research Foundation (JDRF) Artificial Pancreas initiative in 2006. Thus far, we have conducted three closed-loop control clinical trials (totaling 60 subjects with T1D), which demonstrated significantly more time in an acceptable "target" blood glucose range during CLC, and significantly fewer hypoglycemic events during CLC compared to open loop. Our overall objective is to sequentially test, validate, obtain regulatory approval for, and deploy at home, a closed-loop Control-to-Range (CTR) system comprised of two algorithmic components: a Safety Supervision Module (SSM) and an automated Range Correction Module (RCM). The SSM will monitor the safety of the subject's continuous subcutaneous insulin infusion pump (CSII) to prevent hypoglycemia, and will also monitor the integrity of continuous glucose monitor (CGM) data for signal sensor deviations or loss of sensitivity. The RCM will be responsible for the optimal regulation of postprandial hyperglycemic excursions through correction boluses.

The first phase to address our overall objective is a pilot study that will test the ability of a cell-phone-based system to (1) run CTR in an outpatient setting, and (2) be remotely monitored. Specifically, this pilot study entails a hybrid hotel/hospital design targeting adults with T1D that are experienced insulin pump users. Subjects will spend one night in a local hotel, during which the phone-based system will be remotely monitored in an adjacent hotel room for validation that remote system monitoring can successfully occur. Subjects will spend the following day in the hospital, where CTR will be activated, and challenged with meals and a CGM sensor replacement . Subjects will then spend a second night in the hotel for continued evaluation of remote system monitoring, along with outpatient testing of the CTR system run on the phone-based system. This series of admissions will address the first major hurdles that need to be overcome for home deployment of a closed loop CTR system:

Specific Aim 1: The phone-based CTR system can be remotely monitored by nurses/physicians/technicians to confirm appropriate functioning outside of the hospital setting.

Specific Aim 2: The CTR can be deployed outside of the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be aged between 21 (inclusive) and 65 years old. The age of 21 has been chosen because this trial is supported by a US Foundation.
* Patient must have been clinically diagnosed with Type 1 diabetes mellitus. For an individual to be enrolled at least one criterion from each list must be met:

  * Criteria for documented hyperglycemia (at least 1 must be met):

    * Fasting glucose ≥126 mg/dL - confirmed
    * Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥200 mg/dL - confirmed
    * HbA1c ≥6.5% documented - confirmed
    * Random glucose ≥200 mg/dL with symptoms
    * No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes
  * Criteria for requiring insulin at diagnosis (1 must be met):

    * Participant required insulin at diagnosis and continually thereafter
    * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
    * Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
* Use of an insulin pump to treat his/her diabetes for at least 1 year
* Actively using a carbohydrate (CHO) / insulin ratio for insulin bolus adjustments in order to keep blood glucose in a predefined range
* Patient HbA1c is between 6.0% and 9% as measured with DCA2000 or equivalent device
* Patient must demonstrate proper mental status and cognition for the study
* Patient must be willing to avoid consumption of acetaminophen-containing products during the study interventions involving DexCom use
* Patient must be affiliated or beneficiary of a social medical insurance
* Patient has signed informed consent form prior to study entry

Exclusion Criteria:

* Diabetic ketoacidosis within the 6 months prior to enrollment
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
* Pregnancy, breast feeding, or intention of becoming pregnant
* Uncontrolled arterial hypertension (diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg)
* Conditions which may increase the risk of hypoglycemia such as uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation
* History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the DexCom CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
* Anticoagulant therapy other than aspirin
* Oral steroids
* Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admissions.
* Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Known current or recent alcohol or drug abuse
* Medical conditions that would make operating a CGM, cell phone, or insulin pump difficult (e.g. blindness, severe arthritis, immobility)
* Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
* Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥three times the upper reference limit
* Impaired renal function measured as creatinine >1.2 times above the upper limit of normal
* Uncontrolled microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment
* Active gastroparesis requiring current medical therapy
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Uncontrolled thyroid disease
* Known bleeding diathesis or dyscrasia
* Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor
* Unwillingness to withhold dietary supplements two weeks prior to admission and for the duration of the study participation.
* Unwillingness to withhold pramlintide, liraglutide and exenatide for the duration of the study intervention.
* Patient is actively enrolled in another clinical trial or was part of study within 30 days or whose annual study income is over 4 500€
* Persons deprived of freedom, adults protected by law or vulnerable persons

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
estimation of the failure rates of system components | length of admission (hour 42)
  we will estimate the relative frequency of failures (#failures/opportunity of failure) of each following system components: CGM communication (1 failure opportunity every 5min), pump communication (1 failure opportunity every 5min), insulin dose computation (1 failure opportunity every 5min), user interface (1 failure opportunity every 1min).

SECONDARY OUTCOMES:
frequency analysis of lost or inaccurate CGM records | length of admission (42 hours)
  number of CGM data points not received (or corrupted) by the device divided by the total number of possible CGM data points to be received.
percent time of active CTR | length of admission (42h)
  number of minutes the Control-To-Range system was functioning properly (computation of insulin infusion, and insulin actually delivered) divided by the maximum number of minutes the CTR system should have been active (as per protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Avogaro, MD, Principal Investigator — University of Padova Hospital; Boris Kovatchev, PhD, Study Director — University of Virginia
Locations (1):
- Azienda Ospedaliera E Universita Degli Study Di Padova, Padua, Veneto, Italy

REFERENCES:
- [Derived] Kovatchev BP, Renard E, Cobelli C, Zisser HC, Keith-Hynes P, Anderson SM, Brown SA, Chernavvsky DR, Breton MD, Farret A, Pelletier MJ, Place J, Bruttomesso D, Del Favero S, Visentin R, Filippi A, Scotton R, Avogaro A, Doyle FJ 3rd. Feasibility of outpatient fully integrated closed-loop control: first studies of wearable artificial pancreas. Diabetes Care. 2013 Jul;36(7):1851-8. doi: 10.2337/dc12-1965. PMID 23801798